CLINICAL TRIAL: NCT02400307
Title: A Phase 1, Open-Label, Parallel-Group, Adaptive Single-dose Study to Evaluate the Pharmacokinetics of GS-9883 in Subjects With Normal and Impaired Renal Function
Brief Title: Pharmacokinetics of Bictegravir in Adults With Normal and Impaired Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-141-1479; 2015-000898-12 (EudraCT Number)
Record Dates: First submitted 2015-03-17; First posted 2015-03-27 (Estimated); Results first posted 2019-10-11 (Actual); Last update posted 2019-10-11 (Actual); Status verified 2019-09

CONDITIONS: HIV
Keywords: Phase 1; Renally Impaired
MeSH Terms: interventions — bictegravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Severe Renal Impairment (Experimental): Participants with severe renal impairment and matched healthy controls will receive a single dose of bictegravir.
  Interventions: Drug: Bictegravir
- Moderate Renal Impairment (Experimental): Participants with moderate renal impairment and matched healthy controls will receive a single dose of bictegravir.
  Interventions: Drug: Bictegravir
- Mild Renal Impairment (Experimental): Participants with mild renal impairment and matched healthy controls will receive a single dose of bictegravir.
  Interventions: Drug: Bictegravir

INTERVENTIONS:
Drug: Bictegravir — 75 mg tablet administered orally
  Other Names: GS-9883

SUMMARY:
The primary objective of this study is to evaluate the pharmacokinetic (PK) profile of oral bictegravir (formerly GS-9883) in adults with impaired renal function relative to matched, healthy controls with normal renal function. Each participant in the renal impairment groups will be matched for age (± 10 years), gender, and body mass index [BMI (± 20%, 18 ≤ BMI ≤ 40 kg/m^2)] with a participant in the control group.

ELIGIBILITY:
Key Inclusion Criteria:

* All Individuals:

  * Must have a calculated BMI from 18 to 40 kg/m^2, inclusive, at screening
* Individuals with impaired renal function

  * Chronic stable renal impairment without recent clinical change

    * Mild: Creatinine clearance (CrCl) = 60 - 89 mL/min
    * Moderate: CrCl = 30 - 59 mL/min
    * Severe: CrCl = 15 - 29 mL/min
* Healthy individuals

  * CrCl ≥ 90 mL/min

Key Exclusion Criteria:

* All Individuals:

  * Pregnant or lactating females
  * HIV positive or chronic hepatitis B infected
* Individuals with impaired renal function

  * Chronic liver disease
  * Dialysis or anticipated use of dialysis
  * Renal transplant

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-04-17 (Actual); Primary Completion 2015-07-06 (Actual); Study Completion 2015-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (7):
- United States (5):
  - Avail Clinical Research, DeLand, Florida
  - Clinical Pharmacology of Miami, Inc., Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - Prism Clinical Research, Saint Paul, Minnesota
  - New Orleans Center for Clinical Research, Knoxville, Tennessee
- New Zealand (2):
  - Auckland Clinical Studies Limited, Grafton, Auckland
  - Christchurch Clinical Studies Trust, Christchurch

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States and New Zealand. The first participant was screened on 17 April 2015. The last study visit occurred on 13 July 2015.
Pre-assignment Details: 49 participants were screened. No participants were enrolled in the moderate or mild renal impairment adaptive cohorts as a review showed that PK data collected were sufficient to detect any differences between the 2 renal function groups.
Groups:
- Severe Renal Impairment: Participants with severe renal impairment (CrCl = 15 - 29 mL/min) received a single dose of bictegravir 75 mg tablet orally on Day 1 under fed conditions
- Normal Renal Function: Matched healthy control participants with normal renal function (CrCl ≥ 90 mL/min) received a single dose of bictegravir 75 mg tablet orally on Day 1 under fed conditions
Period: Overall Study
Arm/Group | Severe Renal Impairment | Normal Renal Function
Started | 11 | 8
Completed | 10 | 8
Not Completed | 1 | 0
Not completed — Enrolled and Never Dosed | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included participants who received the single dose of bictegravir.
Groups:
- Total: Total of all reporting groups
Arm/Group | Severe Renal Impairment | Normal Renal Function | Total
Number analyzed (Participants) | 10 | 8 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (15.6) | 56 (14.7) | 59 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 7 | 6 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 7 | 6 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 7 | 7 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic (PK) Parameter: AUCinf of Bictegravir (Total)
Description: AUCinf is defined as the area under the plasma concentration versus time curve extrapolated to infinite time.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96, 120 and 144 hours postdose on Day 1
Population: The PK Analysis Set included participants who took the single dose of bictegravir and had at least 1 nonmissing postdose concentration value for bictegravir.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Severe Renal Impairment | Normal Renal Function
Number analyzed (Participants) | 10 | 8
h*ng/mL | 138169.7 (61291.27) | 170105.6 (42213.18)
Statistical Analysis 1: Comparison: Severe Renal Impairment vs Normal Renal Function; A sample size of 8 evaluable participants in each group will provide at least 88% power to reject the null hypothesis that participants with severe impairment have at least 100% increase in bictegravir AUCinf, AUClast, or Cmax compared to participants with normal renal function; Test type: Equivalence — For the power and sample size analysis, it was assumed that a one-sided t-test was performed at an alpha level of 0.05 and the inter-subject standard deviations for the three natural log scale PK parameters are 0.466 or smaller (based on another Gilead study) and the expected difference was 0; Geometric Least-Square Mean (GLSM) Ratio = 72.63, 90% CI 2-sided [48.80 to 108.10]

2. Primary Outcome: PK Parameter: AUCinf of Bictegravir (Free)
Description: Free AUCinf was calculated based on unbound plasma bictegravir (AUCinf × percentage unbound bictegravir ÷ 100 for each participant).
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96, 120 and 144 hours postdose on Day 1
Population: Participants in the PK Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Severe Renal Impairment | Normal Renal Function
Number analyzed (Participants) | 10 | 8
h*ng/mL | 830.6 (266.59) | 824.5 (203.49)
Statistical Analysis 1: Comparison: Severe Renal Impairment vs Normal Renal Function; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; GLSM Ratio = 99.29, 90% CI 2-sided [79.49 to 124.04]

3. Primary Outcome: PK Parameter: AUClast of Bictegravir (Total)
Description: AUClast is defined as the area under the plasma concentration versus time curve from time zero to the last quantifiable concentration.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96, 120 and 144 hours postdose on Day 1
Population: Participants in the PK Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Severe Renal Impairment | Normal Renal Function
Number analyzed (Participants) | 10 | 8
h*ng/mL | 136956.4 (60557.34) | 168876.8 (41706.37)
Statistical Analysis 1: Comparison: Severe Renal Impairment vs Normal Renal Function; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; GLSM Ratio = 72.43, 90% CI 2-sided [48.54 to 108.07]

4. Primary Outcome: PK Parameter: AUClast of Bictegravir (Free)
Description: Free AUClast was calculated based on unbound plasma bictegravir (AUClast × percentage unbound bictegravir ÷ 100 for each participant).
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96, 120 and 144 hours postdose on Day 1
Population: Participants in the PK Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Severe Renal Impairment | Normal Renal Function
Number analyzed (Participants) | 10 | 8
h*ng/mL | 822.5 (263.22) | 818.6 (201.18)
Statistical Analysis 1: Comparison: Severe Renal Impairment vs Normal Renal Function; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; GLSM Ratio = 99.02, 90% CI 2-sided [79.24 to 123.74]

5. Primary Outcome: PK Parameter: Cmax of Bictegravir (Total)
Description: Cmax is defined as the maximum observed plasma concentration of drug.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96, 120 and 144 hours postdose on Day 1
Population: Participants in the PK Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Severe Renal Impairment | Normal Renal Function
Number analyzed (Participants) | 10 | 8
ng/mL | 5977.0 (2079.57) | 7227.5 (2135.56)
Statistical Analysis 1: Comparison: Severe Renal Impairment vs Normal Renal Function; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; GLSM Ratio = 80.32, 90% CI 2-sided [59.56 to 108.30]

6. Primary Outcome: PK Parameter: Cmax of Bictegravir (Free)
Description: Free Cmax was calculated based on unbound plasma bictegravir (Cmax × percentage unbound bictegravir ÷ 100 for each participant).
Time Frame: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72, 96, 120 and 144 hours postdose on Day 1
Population: Participants in the PK Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Severe Renal Impairment | Normal Renal Function
Number analyzed (Participants) | 10 | 8
ng/mL | 37.7 (8.15) | 35.0 (9.94)
Statistical Analysis 1: Comparison: Severe Renal Impairment vs Normal Renal Function; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; GLSM Ratio = 109.80, 90% CI 2-sided [87.46 to 137.85]

7. Secondary Outcome: Percentage of Participants Who Experienced Treatment-Emergent Adverse Events
Description: Treatment-emergent adverse events (TEAEs) are defined as any adverse events (AEs) with an onset date on or after the study drug start date and no later than 30 days after permanent discontinuation of study drug or any AEs leading to premature discontinuation of study drug.
Time Frame: First dose date to Day 31
Population: The Safety Analysis Set included participants who received the single dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Severe Renal Impairment | Normal Renal Function
Number analyzed (Participants) | 10 | 8
percentage of participants | 20.0 | 25.0

8. Secondary Outcome: Percentage of Participants Who Experienced Treatment-Emergent Laboratory Abnormalities
Description: A treatment-emergent graded laboratory abnormality was defined as an increase of at least 1 abnormality grade from the predose assessment and occurring after the predose visit and on or before the date of the administration of study drug plus 30 days. The most severe graded abnormality from all tests was counted for each participant. Toxicity grade was defined as follows: Grade 1 = Mild, Grade 2 = Moderate, Grade 3 = Severe, and Grade 4 = Life-threatening.
Time Frame: First dose date to Day 31
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Severe Renal Impairment | Normal Renal Function
Number analyzed (Participants) | 10 | 8
percentage of participants
  Grade 1 | 20.0 | 25.0
  Grade 2 | 40.0 | 25.0
  Grade 3 | 40.0 | 0
  Grade 4 | 0 | 0

ADVERSE EVENTS:
Time Frame: First dose date to Day 31
Description: The Safety Analysis Set included participants who received the single dose of bictegravir.
Arm/Group | Severe Renal Impairment | Normal Renal Function
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/8
Other Adverse Events (participants affected / at risk) | 2/10 | 2/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Severe Renal Impairment (N=10) | Normal Renal Function (N=8)
Constipation (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years